CLINICAL TRIAL: NCT03390491
Title: OnTrack>An Online Role-Playing Game for Young People With First Episode Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Social Innovation, Massachusetts (Other)
Collaborators: Research Foundation for Mental Hygiene, Inc. (Other); New York State Psychiatric Institute (Other); University of Maryland, College Park (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: #7643; 2R44MH105013-02 (NIH)
Record Dates: First submitted 2017-12-19; First posted 2018-01-04 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Psychosis; Schizoaffective Disorder; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OnTrack>TheGame (OTG) (Experimental): Participants randomized to the OTG group (n=100) will have the option to play the online role-playing game for a period of 2 months. They will receive weekly email reminders that the game remains available to them.
  Interventions: Behavioral: OnTrack>TheGame (OTG)
- Recovery Videos (RV) (Other): Participants randomized to the RV group (n=100) will have the option to visit a website that will contain the recovery videos and the static information that is contained in the game. The RV group will also have 2 months to view the materials on the website and will receive weekly email reminders that the website/videos remain available to them. At the end of the study (after the follow-up assessment), the RV participants will be provided access to the game.
  Interventions: Behavioral: Recovery Videos (RV)

INTERVENTIONS:
Behavioral: OnTrack>TheGame (OTG) — OTG clients will be informed that the game can be played on a computer or a tablet and the time estimate for completing the game is approximately 5-8 hours. OnTrack>The Game offers players the opportunity to immerse in a fictional neighborhood that centers around four domains for supportive recovery as defined by SAMHSA: health, home, purpose and community. The player interacts with other game characters including new acquaintances, friends/peers, a family member, and a treatment team, allowing the player to practice social and communication skills, while fostering personal relationships and building a support network. Additionally, the game provides players with helpful resources including psychoeducation materials and videos of real people who have experienced a first episode of psychosis, sharing their stories of hope and recovery. As a whole, the game provides a safe environment to promote goal attainment and recovery.
  Arms: OnTrack>TheGame (OTG)
Behavioral: Recovery Videos (RV) — As described, RV clients will have access to a website that includes recovery videos and static psychoeducation materials. In this condition, mental health providers will also ask about possible reactions to viewing the recovery videos and information on the website.
  Arms: Recovery Videos (RV)

SUMMARY:
The research team will develop and test a prototype version of OnTrack>An Online Role-Playing Game (OnTrack>The Game or OTG), an online role-playing game designed for youth and young adults experiencing First Episode Psychosis (FEP). Phase I showed positive changes in quantitative measures of hope and recovery, as well as an enthusiastic response to the prototype as evidenced by qualitative interviews. In Phase II, the research team will refine, expand and finalize OTG and evaluate the effectiveness of OTG.

DETAILED DESCRIPTION:
The proposed mixed-methods Phase II study will use standardized measures and semi-structured qualitative interviews to achieve the following aims:

1. Product aim: To refine, expand, and finalize OnTrack>The Game. Building on the Phase I prototype, the investigators will improve functionality, expand the play spaces and levels, add interaction with non-player characters, include more resources on FEP, and expand the library of videos on hope and recovery.
2. Primary research aim: To evaluate the effectiveness of a role-playing game (OTG) in increasing empowerment, decreasing stigma concerns, and improving treatment engagement.

   Hypothesis 1: Compared to control condition (Recovery Videos, or RV), participants in OTG will report significantly increased empowerment at 2 months post-intervention compared to baseline.

   Hypothesis 2: Compared to the control condition (RV), participants randomized to the OTG condition will report significantly increased empowerment, decreased stigma concerns, and greater treatment engagement at the 5-month follow-up compared to baseline.
3. Secondary research aim: To determine if changes in empowerment and stigma concerns mediate the effect of OnTrack>The Game on treatment engagement.

Hypothesis 3: Increases in hope, attitudes toward treatment, and self-efficacy and decreases in stigma concerns at post treatment will partially mediate the improvement in treatment engagement at follow-up.

Approach

Overview and Rationalization of Study Design: Phase II is a randomized controlled trial (RCT) enrolling 200 clients randomized to OTG or a control condition of RVs in a 1:1 ratio. The investigators will recruit these participants from OnTrackNY's Early Intervention for Psychosis (EIP) clinical centers after screening for eligibility. After consent and Baseline data collection, participants will be randomly assigned to either OTG or RV, which will be available to them for two months. Following an intent-to-treat framework, the investigators will then assess each client participant at 2 additional time points regardless of participation in their assigned condition: post-intervention (immediately after the 2 month intervention has completed), then follow-up at 3 months post-intervention.

Ten clinicians working with these clients will also be recruited for semi-structured key informant qualitative interviews. Twenty client interviews will also be conducted, 10 from each condition. The investigators' rationale for selecting a randomized controlled design stems from Phase I findings, which suggest that the game may be effective in addressing young people's hopefulness, stigma, and understanding around first episode psychosis. An RCT design will allow the research team to examine how specific aspects of the game impact outcomes in these areas, as compared to more static, passive online resource.

Study Setting: OnTrackNY is New York State's coordinated specialty care (CSC) program. Funded by state dollars, a SAMHSA Health Transitions Grant, and Mental Health Block Grant funds, the state currently supports 13 teams throughout the state. Eight additional programs are expected to come on line within the next 6 months. The program serves young adults ages 16 to 30. To date, a total of 290 individuals have been enrolled. Across the sites, clients are 69% male; mean age of 21; 19% are under the age of 18; racial/ethnic breakdown is as follows: 42% White, 39% Black, 10% Asian, 9% Other, and 23% Hispanic.

ELIGIBILITY:
Inclusion Criteria:

Client inclusion criteria:

* Currently enrolled in OnTrackNY
* English speaking
* Clinically stable (not in crisis or experiencing severe or elevated symptoms)
* Capable of providing informed consent
* Regular access to a computer or tablet (at home or at their OnTrack site)
* Working email address and access to email
* Enrolled in OnTrackNY less than 19 months
* Parent or guardian permission for minors (age 16-17)

Exclusion Criteria for Clients:

• Not meeting inclusion criteria. No other exclusion criteria.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Treatment Engagement | At time point 3 (five months after baseline)
  Improved treatment engagement in participants from OTG condition compared to the control condition, RV (measured by a. Signh O'Brien Level of Engagement Scale, b. Engagement with CSC program determined by record review)
Empowerment | at time point 2 (two months after baseline); and at time point 3 (five months after baseline)
  Increased empowerment in participants from OTG condition compared to the control condition, RV (measured by: a. Herth Hope Index, b. Recovery Attitude Questionnaire, c. Roger's Empowerment Scale)
Stigma | at time point 3 (five months after baseline)
  Decreased stigma concerns in participants from OTG condition compared to the control condition, RV (measured by a. Questionnaire on Anticipated Stigma, b. Rüsch Stigma Stress)

SECONDARY OUTCOMES:
Empowerment and Stigma Mediating Effect on Treatment Engagement | do increases in empowerment and decreases in stigma concerns at time point 2 (2 months after baseline), mediate the effect of OTG on treatment engagement at time point 3 (5 months after baseline)
  Do increases in empowerment and decreases in stigma concerns mediate the effect of OTG on treatment engagement

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Marcogliese, PhD, Principal Investigator — Center for Social Innovation
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dixon LB, Goldman HH, Bennett ME, Wang Y, McNamara KA, Mendon SJ, Goldstein AB, Choi CW, Lee RJ, Lieberman JA, Essock SM. Implementing Coordinated Specialty Care for Early Psychosis: The RAISE Connection Program. Psychiatr Serv. 2015 Jul;66(7):691-8. doi: 10.1176/appi.ps.201400281. Epub 2015 Mar 16. PMID 25772764
- [Background] Kane JM, Robinson DG, Schooler NR, Mueser KT, Penn DL, Rosenheck RA, Addington J, Brunette MF, Correll CU, Estroff SE, Marcy P, Robinson J, Meyer-Kalos PS, Gottlieb JD, Glynn SM, Lynde DW, Pipes R, Kurian BT, Miller AL, Azrin ST, Goldstein AB, Severe JB, Lin H, Sint KJ, John M, Heinssen RK. Comprehensive Versus Usual Community Care for First-Episode Psychosis: 2-Year Outcomes From the NIMH RAISE Early Treatment Program. Am J Psychiatry. 2016 Apr 1;173(4):362-72. doi: 10.1176/appi.ajp.2015.15050632. Epub 2015 Oct 20. PMID 26481174
- [Background] Abdel-Baki A, Lal S, D-Charron O, Stip E, Kara N. Understanding access and use of technology among youth with first-episode psychosis to inform the development of technology-enabled therapeutic interventions. Early Interv Psychiatry. 2017 Feb;11(1):72-76. doi: 10.1111/eip.12250. Epub 2015 May 22. PMID 26011657
- [Background] Mohr DC, Burns MN, Schueller SM, Clarke G, Klinkman M. Behavioral intervention technologies: evidence review and recommendations for future research in mental health. Gen Hosp Psychiatry. 2013 Jul-Aug;35(4):332-8. doi: 10.1016/j.genhosppsych.2013.03.008. Epub 2013 May 8. PMID 23664503
- [Background] Shandley K, Austin D, Klein B, Kyrios M. An evaluation of 'Reach Out Central': an online gaming program for supporting the mental health of young people. Health Educ Res. 2010 Aug;25(4):563-74. doi: 10.1093/her/cyq002. Epub 2010 Feb 11. PMID 20150530
- [Background] Lieberman JA, Dixon LB, Goldman HH. Early detection and intervention in schizophrenia: a new therapeutic model. JAMA. 2013 Aug 21;310(7):689-90. doi: 10.1001/jama.2013.8804. No abstract available. PMID 23989167
- [Background] Stroup, T. S., Lawrence, R. E., Abbas, A. I., Miller, B. R., Perkins, D. O., Lieberman J. A. (2013). Schizophrenia spectrum and other psychotic disorders. In: R. E. Hales, S. C. Yudofsky, & L. Roberts (Eds.). The American psychiatric publishing textbook of psychiatry (6th ed.). Washington, DC: American Psychiatric Publishing.
- [Background] Wu EQ, Birnbaum HG, Shi L, Ball DE, Kessler RC, Moulis M, Aggarwal J. The economic burden of schizophrenia in the United States in 2002. J Clin Psychiatry. 2005 Sep;66(9):1122-9. doi: 10.4088/jcp.v66n0906. PMID 16187769
- [Background] Baranowski T, Buday R, Thompson DI, Baranowski J. Playing for real: video games and stories for health-related behavior change. Am J Prev Med. 2008 Jan;34(1):74-82. doi: 10.1016/j.amepre.2007.09.027. PMID 18083454
- [Background] Hieftje K, Edelman EJ, Camenga DR, Fiellin LE. Electronic media-based health interventions promoting behavior change in youth: a systematic review. JAMA Pediatr. 2013 Jun;167(6):574-80. doi: 10.1001/jamapediatrics.2013.1095. PMID 23568703
- [Background] Armstrong S. Video games on prescription. BMJ. 2014 Sep 15;349:g5615. doi: 10.1136/bmj.g5615. No abstract available. PMID 25224744
- [Background] Jones CM, Scholes L, Johnson D, Katsikitis M, Carras MC. Gaming well: links between videogames and flourishing mental health. Front Psychol. 2014 Mar 31;5:260. doi: 10.3389/fpsyg.2014.00260. eCollection 2014. PMID 24744743
- [Background] Perkins DO, Gu H, Boteva K, Lieberman JA. Relationship between duration of untreated psychosis and outcome in first-episode schizophrenia: a critical review and meta-analysis. Am J Psychiatry. 2005 Oct;162(10):1785-804. doi: 10.1176/appi.ajp.162.10.1785. PMID 16199825
- [Background] Agarkar S. A case of prolonged duration of untreated psychosis: barriers to treatment and strategies to improve the outcome. Clin Schizophr Relat Psychoses. 2012 Apr;6(1):45-8. PMID 22453869
- [Background] Bottlender R, Sato T, Jager M, Wegener U, Wittmann J, Strauss A, Moller HJ. The impact of the duration of untreated psychosis prior to first psychiatric admission on the 15-year outcome in schizophrenia. Schizophr Res. 2003 Jul 1;62(1-2):37-44. doi: 10.1016/s0920-9964(02)00348-1. PMID 12765741
- [Background] Goh, D. H., Ang, R. P., & Tan, H. C. (2008). Strategies for designing effective psychotherapeutic gaming interventions for children and adolescents. Computers in Human Behavior, 24(5), 2217-2235.
- [Background] Wilkinson N, Ang RP, Goh DH. Online video game therapy for mental health concerns: a review. Int J Soc Psychiatry. 2008 Jul;54(4):370-82. doi: 10.1177/0020764008091659. PMID 18720897
- [Background] Batson, L., & Feinberg, S. (2006). Game designs that enhance motivation and learning for teenagers. Electronic Journal for the Integration of Technology in Education, 5(1), 34-43.
- [Background] Neal, J.W., Neal, Z.P., VanDyke, E., & Kornbluh, M. (2015). Expediting the analysis of qualitative data in evaluation: A procedure for the Rapid Identification of Themes From Audio Recordings (RITA). American Journal of Evaluation, 36(1), 118-132. doi: 10.1177/1098214014536601
- [Background] Rusch N, Corrigan PW, Wassel A, Michaels P, Olschewski M, Wilkniss S, Batia K. A stress-coping model of mental illness stigma: I. Predictors of cognitive stress appraisal. Schizophr Res. 2009 May;110(1-3):59-64. doi: 10.1016/j.schres.2009.01.006. Epub 2009 Mar 6. PMID 19269140
- [Background] Herth K. Abbreviated instrument to measure hope: development and psychometric evaluation. J Adv Nurs. 1992 Oct;17(10):1251-9. doi: 10.1111/j.1365-2648.1992.tb01843.x. PMID 1430629
- [Background] Rogers ES, Chamberlin J, Ellison ML, Crean T. A consumer-constructed scale to measure empowerment among users of mental health services. Psychiatr Serv. 1997 Aug;48(8):1042-7. doi: 10.1176/ps.48.8.1042. PMID 9255837
- [Background] Gabbidon J, Brohan E, Clement S, Henderson RC, Thornicroft G; MIRIAD Study Group. The development and validation of the Questionnaire on Anticipated Discrimination (QUAD). BMC Psychiatry. 2013 Nov 7;13:297. doi: 10.1186/1471-244X-13-297. PMID 24199691
- [Background] Shortreed SM, Laber E, Scott Stroup T, Pineau J, Murphy SA. A multiple imputation strategy for sequential multiple assignment randomized trials. Stat Med. 2014 Oct 30;33(24):4202-14. doi: 10.1002/sim.6223. Epub 2014 Jun 11. PMID 24919867
- [Derived] Jankowski S, Ferreira K, Mascayano F, Donovan E, Rahim R, Birnbaum ML, Yum-Chan S, Medoff D, Marcogliese B, Fang L, Nicholson T, Dixon L. A Serious Game for Young People With First Episode Psychosis (OnTrack>The Game): Qualitative Findings of a Randomized Controlled Trial. JMIR Ment Health. 2022 Apr 6;9(4):e33526. doi: 10.2196/33526. PMID 35384847
- [Derived] Roberts MT, Lloyd J, Valimaki M, Ho GW, Freemantle M, Bekefi AZ. Video games for people with schizophrenia. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD012844. doi: 10.1002/14651858.CD012844.pub2. PMID 33539561